CLINICAL TRIAL: NCT00000894
Title: Ganciclovir-Cidofovir CMV Retinitis Trial (GCCRT)
Brief Title: Comparison of Two Drugs, Cidofovir and Ganciclovir, in Treating Patients With AIDS Who Have CMV Retinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 350
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-02-23 (Estimated); Status verified 2003-06

CONDITIONS: Cytomegalovirus Retinitis; HIV Infections
Keywords: Infusions, Intravenous; Ganciclovir; Drug Therapy, Combination; Administration, Oral; Antiviral Agents; Drug Implants; Cytomegalovirus Retinitis; Eye; cidofovir
MeSH Terms: conditions — Cytomegalovirus Retinitis; HIV Infections; Multiple Acyl Coenzyme A Dehydrogenase Deficiency | interventions — Cidofovir; Probenecid; Ganciclovir

INTERVENTIONS:
Drug: Cidofovir
Drug: Probenecid
Drug: Ganciclovir

SUMMARY:
To compare cidofovir with a commonly used treatment regimen, ganciclovir given by mouth (oral) and through an eye device (intraocular) , in order to determine the safety and effectiveness of cidofovir in preventing vision loss in patients who have AIDS complicated by CMV (cytomegalovirus) retinitis.

Cidofovir needs to be compared to ganciclovir to determine the best way to treat CMV retinitis.

DETAILED DESCRIPTION:
While cidofovir is effective in suppressing retinitis and prolonging time to progression, no studies have compared cidofovir to other therapies and its place in the treatment of CMV retinitis remains unexplored. By combining the ganciclovir intraocular device (slows retinitis progression) with oral ganciclovir (has the potential to treat both the ocular disease and to suppress dissemination to the contralateral eye and the viscera), without the use of a central venous catheter, this combination has become increasingly common. For these reasons, a comparative trial of cidofovir to other therapies is appropriate.

After being stratified by the clinic and by stage of disease, patients are randomized to 1 of 2 treatment arms: intravenous (IV) cidofovir (Group I) or intraocular ganciclovir device plus oral ganciclovir (Group II). Group I: Cidofovir is administered IV once weekly for 2 consecutive weeks, then every 2 weeks thereafter. If progression occurs, oral ganciclovir is added to treatment or if this regimen is not tolerated, patients are treated according to the best medical judgment. Concurrent oral probenecid and intravenous hydration are administered with each cidofovir infusion. Group II: An intraocular ganciclovir device is surgically implanted at baseline and then every 6 to 8 months and ganciclovir is administered orally. If more than 1 progression or unacceptable toxicity occurs, patients are treated according to the best medical judgment.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are 13 years of age or older (parent or guardian consent required if under 18).
* Agree to practice sexual abstinence or use effective birth control during and for 90 days after the study.
* Have AIDS.
* Have CMV retinitis.

Exclusion Criteria

You will not be eligible for this study if you:

* Have a history of heart or kidney disease.
* Have medical problems which would prevent you from completing the study.
* Are pregnant.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300
Dates: Primary Completion 2000-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Univ of Southern California / LA County USC Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Univ of Miami / Bascom Palmer Eye Institute, Miami, Florida
  - Emory Eye Clinic, Atlanta, Georgia
  - Northwestern Univ / SOCA, Chicago, Illinois
  - Charity Hosp / Tulane Univ Med School, New Orleans, Louisiana
  - Johns Hopkins Hosp, Baltimore, Maryland
  - Cornell Univ Med Ctr, New York, New York
  - New York Hosp / Cornell Med Ctr, New York, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Texas Galveston, Galveston, Texas